CLINICAL TRIAL: NCT01184560
Title: A Randomized, Double-blind, Placebo-controlled, Investigator-initiated Study to Assess the Additional Weight Loss Effect of Orlistat Used in Combination With Sibutramine
Brief Title: Assess the Additional Weight Loss Effect of Orlistat Used in Combination With Sibutramine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Kyoungkon Kim/Principal Investigator, GachonGill Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-OPS
Record Dates: First submitted 2010-08-16; First posted 2010-08-19 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2009-10

CONDITIONS: Obesity
Keywords: obesity
MeSH Terms: conditions — Obesity | interventions — sibutramine; Orlistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sibutramine + Orlistat (Experimental): A lipase inhibitor used for weight loss. Lipase is an enzyme found in the bowel that assists in lipid absorption by the body. Orlistat blocks this enzyme, reducing the amount of fat the body absorbs by about 30%. It is known as a "fat blocker". Because more oily fat is left in the bowel to be excreted, Orlistat can cause an oily anal leakage and fecal incontinence
  Interventions: Drug: Sibutramine; Drug: Orlistat
- Sibutramine + Orlistat(Placebo) (Placebo Comparator): 1. Sibutramine : one of components included into Diet Pills. This reduces appetite, normalizes amount of cholesterol in blood, and reduces abdominal fat.
  2. Orlistat : A lipase inhibitor used for weight loss. Lipase is an enzyme found in the bowel that assists in lipid absorption by the body. Orlistat blocks this enzyme, reducing the amount of fat the body absorbs by about 30%. It is known as a "fat blocker". Because more oily fat is left in the bowel to be excreted, Orlistat can cause an oily anal leakage and fecal incontinence.
  Interventions: Drug: Sibutramine; Drug: Orlistat

INTERVENTIONS:
Drug: Sibutramine — ○ Dosing standard Run-in period: All subjects would administer Sibutramine placebo 1 capsule (once daily) and Orlistat placebo 1 capsule (three times daily). The total dosing period is 2 weeks.
  Treatment period: The total dosing period is 12 weeks.
  * Sibutramine monotherapy group: Sibutramine 1 capsule once daily + Orlistat placebo 1 capsule three times daily
  * Orlistat and Sibutramine combination group: Sibutramine 1 capsule once daily + Orlistat 1 capsule three times daily
Drug: Orlistat — ○ Dosing standard Run-in period: All subjects would administer Sibutramine placebo 1 capsule (once daily) and Orlistat placebo 1 capsule (three times daily). The total dosing period is 2 weeks.
  Treatment period: The total dosing period is 12 weeks.
  * Sibutramine monotherapy group: Sibutramine 1 capsule once daily + Orlistat placebo 1 capsule three times daily
  * Orlistat and Sibutramine combination group: Sibutramine 1 capsule once daily + Orlistat 1 capsule three times daily

SUMMARY:
The purpose of this study, conducted academic Pilot research purposes, this is not clear as to permit. when orlistat to sibutramine merge if there are additional effects of BMI and group, which has an attribute that is greater for the combined effect is to analyze.

* Study phase: Investigator-initiated clinical study (Pilot study)
* Method of blinding: Double-blind
* Control: Placebo-controlled
* Assignment method: Randomization (Sibutramine monotherapy group: Orlistat and Sibutramine combination group = 1 : 1)
* Studied disease: Obesity
* Study population: Subjects eligible for inclusion/exclusion criteria
* Dosing period: Total 18 weeks Run-in period (2 weeks), dosing period (12 weeks) and post-dosing observation period (4 weeks)

DETAILED DESCRIPTION:
After the screening period, patients eligible for inclusion/exclusion criteria would administer Sibutramine placebo and Orlistat placebo during 2 weeks of the run-in period, Subsequently, subjects are randomized to 2 groups of the Sibutramine monotherapy group and the Orlistat and Sibutramine combination group. Sibutramine monotherapy group would receive Sibutramine 10mg once daily and Orlistat placebo three times daily for 12 weeks; the Orlistat and Sibutramine combination group would receive Sibutramine 10mg once daily and Orlistat 120mg three times daily for 12 weeks. After completing the dosing period, the occurrence of adverse events would be checked for 4 weeks and the study would be completed.

Body weight, abdominal CT(Computed Tomography)(visceral fat examination), body fat analysis, etc. would be measured before the study initiation and after 14 weeks of treatment, and comparatively analyzed. A two sample t-test is conducted for the inter-group comparison and a paired t-rest is conducted for the comparison between baseline and after 14 weeks after the study initiation.

ELIGIBILITY:
MAOInclusion Criteria:

1. A patient who gave one's voluntary written consent to participate in this clinical study
2. Aged ≥ 18 and < 50 years old
3. An obese patient with a body mass index (BMI) ≥ 27 kg/m2
4. In case of a women, premenopausal woman

Exclusion Criteria:

1. A patient with the weight change ≥ 5% over the past 3 months
2. A patient who was receiving a MAO(monoamine oxldase) inhibitor within 1 months of screening
3. A patient with an active acute or chronic disease at the participation of the study
4. A patient with the malignancy history within the past 5 years
5. A patient diagnosed with secondary obesity (Cushing's syndrome, thyroid disease, etc.)
6. A patient with a significant cardiovascular disease (coronary vascular disease, congestive heart failure, peripheral arterial obstructive disease, arrhythmia, cerebrovascular disease, etc.), poorly controlled hypertension defined by JNC(Joint National Committee) 7 guidelines, diabetes, severe hepatic/renal disease and CNS(Central Nervous System) disease, drug abuse, psychiatric disorder, positive prostatic hyperplasia concurrent with urinary retention and glaucoma within the past 1 year according to medical records
7. A patient falling under the followings from screening test results Hemoglobin < 10g/L or platelets < 100* 103/μL Total bilirubin > 2.0mg/dL Serum GOT(Glutamate oxaloacetate transaminase) or GPT(glutamic pyruvate transaminase) > 120 IU/L Serum creatinine > 1.4mg/dL Serum uric acid > 10mg/dL Thyroid stimulating hormone < 0.1μIU/mL or > 6.5 μIU/mL
8. A patient with clear unexplained abnormal findings in chest X-ray, urinalysis, electrocardiogram
9. A pregnant women or breastfeeding mother
10. A patient participating in another clinical study other than this study
11. Other patient who is legally and mentally not appropriate to participate in a clinical study, at the judgment of the investigator
12. A person who participated in other clinical study within the past 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Weight | with in 18weeks
  Weight
BMI(Body Mass Index) | with in 18weeks
  BMI(Body Mass Index)
waist circumference | with in 18weeks
  waist circumference
blood pressure | with in 18weeks
  blood pressure
fat mass | with in 18weeks
  fat mass
visceral fat mass improvement | with in 18weeks
  visceral fat mass improvement

SECONDARY OUTCOMES:
Lipid profile | with in 18weeks
  Total cholesterol, HDL-C(high-density lipoprotein-cholesterol), LDL-C(low-density lipoprotein-cholesterol), Triglyceride improvement
Adipokines improvement | with in 18weeks
  Serum insulin, adiponectin, leptin, ghrelin, serum ostecalcin, urine deoxypyridinolin

CONTACTS AND LOCATIONS:
Overall Officials: Kim Kyoungkon, Principal Investigator — GachonGill Medical Center
Locations (1):
- GachonGill Medical Center, Inchon, Namdong-gu, South Korea

REFERENCES:
- [Derived] Ko KD, Kim KK, Suh HS, Hwang IC. Associations between the GNB3 C825T polymorphism and obesity-related metabolic risk factors in Korean obese women. J Endocrinol Invest. 2014 Nov;37(11):1117-20. doi: 10.1007/s40618-014-0182-6. Epub 2014 Oct 4. PMID 25280441
- [Derived] Kim KK, Suh HS, Hwang IC, Ko KD. Influence of eating behaviors on short-term weight loss by orlistat and anorectic agent. Eat Behav. 2014 Jan;15(1):87-90. doi: 10.1016/j.eatbeh.2013.10.019. Epub 2013 Oct 31. PMID 24411757
- [Derived] Hwang IC, Park JY, Ahn HY, Kim KK, Suh HS, Ko KD, Kim KA. Effects of CYP3A5, CYP2C19, and CYP2B6 on the clinical efficacy and adverse outcomes of sibutramine therapy: a crucial role for the CYP2B6*6 allele. Clin Chim Acta. 2014 Jan 20;428:77-81. doi: 10.1016/j.cca.2013.11.007. Epub 2013 Nov 19. PMID 24262967
- [Derived] Hwang IC, Kim KK, Ahn HY, Suh HS, Oh SW. Effect of the G-protein beta3 subunit 825T allele on the change of body adiposity in obese female. Diabetes Obes Metab. 2013 Mar;15(3):284-6. doi: 10.1111/dom.12023. Epub 2012 Nov 8. PMID 23061407